CLINICAL TRIAL: NCT00199277
Title: Randomized, Parallel Group, Clinical Trial Comparing Intravenous Iron Sucrose Versus Oral Ferrous Sulphate in the Treatment of Perioperative Iron Deficiency in Patients With Colo-Rectal Neoplasm and Iron Deficiency Anemia.
Brief Title: Iron Therapy in Colo-Rectal Neoplasm and Iron Deficiency Anemia: Intravenous Iron Sucrose Versus Oral Ferrous Sulphate.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: J. Uriach and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM01VEN/4/03
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Colorectal Neoplasm; Iron Deficiency Anemia
MeSH Terms: conditions — Colorectal Neoplasms; Anemia, Iron-Deficiency | interventions — Iron

INTERVENTIONS:
Drug: i.v. iron sucrose
Drug: Oral iron

SUMMARY:
The main objective of this study is to evaluate the efficacy of intravenous iron sucrose in increasing preoperative haemoglobin values in patients with colo-rectal neoplasm and iron deficiency anemia, compared to the standard treatment with oral iron. It will also determine whether intravenous iron sucrose administration improves outcomes such as postoperative haemoglobin values, serum ferritin values, transfusional needs, postoperative complications, or length of hospital stay.

DETAILED DESCRIPTION:
Most patients with colorectal neoplasm have iron deficiency, which can be triggered in the pre-operative period by a decrease of iron intake and the bleeding in the site of neoplasm.

In the postoperative period, iron deficiency can be aggravated by surgical bleeding.

Iron plays a leading rol in haemoglobin production, cell mitosis and immune system. Animal experimentation has shown that induced iron deficiency and mild anemia lead to postoperative mortality and lactacidemia in a model of peritonitis.

Moreover, anemia is the main risk factor to require intra and postoperative blood transfusions, and iron deficiency and anemia are associated to a larger number of postoperative complications (infections and longer hospital stay).

Oral iron therapy is the standard treatment in patients with preoperative iron deficiency, but iron levels inside red cells may not reach normality in time before surgery, and it can not be resumed until the patient can start again oral feeding.

In these patients, any increase in preoperative haemoglobin decreases the risk to need a blood transfusion during or after surgery.

This trial will compare standard oral iron and intravenous iron.

ELIGIBILITY:
Inclusion Criteria:

* Non-recurrent colorectal neoplasm, surgically resectable
* Anemia

Exclusion Criteria:

* Severe renal impairment
* High anesthetic risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150

PRIMARY OUTCOMES:
Preoperative variations in hemoglobin.

SECONDARY OUTCOMES:
Postoperative variations in hemoglobin.
Blood transfusion needs (pre, intra and postoperative)
Postoperative complications:
- Pulmonary thromboembolism
- Infections
- Reintervention
- Death
Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Pere Poch Martí, MD, Study Chair — Fundació Hospital-Asil de Granollers (Barcelona, Spain)
Locations (5):
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Comarcal Sant Jaume de Calella., Calella, Barcelona
  - Fundació Hospital Asil de Granollers, Granollers, Barcelona
  - Consorci Sanitari del Maresme, Mataró, Barcelona
  - Hospital Miguel Servet, Zaragoza, Zaragoza